CLINICAL TRIAL: NCT04070235
Title: A Multicenter, Open-Label Study to Evaluate the Efficacy and Safety of SH229 Tablets Combined With Daclatasvir Dihydrochloride Tablets in Treatment Adult Patients With Chronic Hepatitis C
Brief Title: SH229 Tablets Combined With Daclatasvir Dihydrochloride Tablets in Treatment Adult Patients With Chronic Hepatitis C
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nanjing Sanhome Pharmaceutical, Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHC005-II/III-01
Record Dates: First submitted 2019-08-11; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C virus; SH229
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — daclatasvir

STUDY DESIGN:
Intervention Model Description: Phase 2 is parallel;Phase 3 is single group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- SH229/DCV 400mg/60mg (Experimental): HCV GT 1-6 participants were medicated with SH229 tablets 400 mg once daily and DCV tablets 60 mg once daily QD (n=40) for 12weeks
  Interventions: Drug: SH229 tablets; Drug: Daclatasvir dihydrochloride
- SH229/DCV 600mg/60mg (Experimental): HCV GT 1-6 participants were medicated with SH229 tablets 600 mg once daily and DCV tablets 60 mg once daily (n=40).
  Interventions: Drug: SH229 tablets; Drug: Daclatasvir dihydrochloride
- SH229/DCV 800mg/60mg (Experimental): HCV GT 1-6 participants were medicated with SH229 tablets 800 mg once daily and DCV tablets 60 mg once daily (n=40).
  Interventions: Drug: SH229 tablets; Drug: Daclatasvir dihydrochloride
- SH229/DCV (Experimental): HCV GT 1-6 participants were medicated with SH229 tablets 400 mg,600 mg or 800 mg once daily and DCV tablets 60 mg once daily
  Interventions: Drug: SH229 tablets; Drug: Daclatasvir dihydrochloride

INTERVENTIONS:
Drug: SH229 tablets — SH229 400 mg was provided in 4 tablets, 100mg each；SH229 600 mg was provided in 6 tablets , 100mg each；SH229 800 mg in was provided in 8tablets , 100mg each。
  Other Names: Holybuvir
Drug: Daclatasvir dihydrochloride — Daclatasvir dihydrochloride was provided in a single tablet of 60 mg.
  Other Names: DAKLINZA

SUMMARY:
Phase II: Exploring the efficacy and safety of different doses of SH229 tablets combined with fixed-dose Daclatasvi dihydrochloride (DCV) tablets in the treatment of adult patients with chronic hepatitis C for 12 weeks, providing a basis for the design and implementation of phase III clinical trials.

Phase III: Confirmation of the efficacy and safety of SH229 tablets combined with Daclatasvi dihydrochloride (DCV) tablets in the treatment of adult patients with chronic hepatitis C for 12 weeks, providing a sufficient basis for drug registration and clinical use.

DETAILED DESCRIPTION:
It is estimated that China has a population of over 10 million infected with HCV and also a highly variable HCV genotype geographic distribution. A simple, universal, non-genotype-specific treatment regimen is preferred for anti-HCV treatment in clinical practice and public health. The combination regimen of SH229 and DCV is expected to completely suppress HCV replication in subjects chronically infected with HCV and achieve a sustained virologic response.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent.
* Subjects should be able to follow the instructions for the study drug and be able to complete screening, on-treatment, and post treatment assessments.
* Male or female, age above 18 years
* Body mass index ( BMI ) between 18 and 32 kg/m2 at Screening.
* Confirmation of chronic HCV infection, which meets one of the following: (a) positive for anti-HCV antibodies, HCV RNA or HCV genotyping results within ≤ 6 months of screening, or (b) liver biopsy ≤ 12 months of screening.
* HCV RNA above 10^4 IU/mL at Screening by the Central Laboratory.
* HCV genotype 1, 2, 4, 5, 6, or indeterminate assessed at Screening by the Central Laboratory.
* Classification as treatment naïve or treatment experienced (approximately 20% of subjects may be treatment experienced):

  1. Treatment naïve is defined as having never been exposed to approved or experimental HCV-specific direct-acting antiviral agents ( DAA ) or prior treatment of HCV with interferon either with or without RBV.
  2. Treatment experienced is defined as prior treatment failure to a regimen containing IFN-based antiviral (INF-α, β or PEG-IFN ± ribavirin) and met one of the following: (i) Non-Responder: Subject did not achieve undetectable HCV RNA levels while ontreatment,, (ii) Relapse/Breakthrough: Subject achieved undetectable HCV RNA levels duringtreatment but did not achieve SVR, (iii) Terminate the treatment , according to associated-HCV therapy adverse events by subject reported or medical records demonstrated.
* Cirrhosis Determination (approximately 20% of subjects may have cirrhosis)：

  1. Cirrhosis is defined as any one of the following: (i) Fibroscan with a result of >12.5 kPa within ≤ 6 months of screening, (ii) Liver biopsy showing cirrhosis within ≤ 12 months of screening.
  2. Absence of cirrhosis is defined as any one of the following:(i) Fibroscan with a result of ≤ 12.5 kPa within ≤ 6 months of screening, (ii) Liver biopsy showing non-cirrhosis within ≤ 12 months of screening.

Exclusion Criteria:

* Exposure nucleotide analogue including HCV NS3-4A inhibitor, HCV NS5B inhibitor or any HCV NS5A inhibitor before baseline/Day 1.
* Receive IFN-based antiviral therapy within 6 months prior to baseline/day 1.
* Oral or injection of RBV within 3 months prior to baseline/Day 1.
* Systemic use of potent immunomodulators (eg, adrenocortical hormone, thymosin alpha, etc.) for more than 2 weeks prior to baseline/day 1, or expected to be exposed to these agents during the study.
* Use of amiodarone within 2 months before baseline/day 1.
* Positive for Hepatitis B surface antigen (HBsAg) or anti-human immunodeficiency virus antibody (HIV Ab) at screening.
* Evidence of decompensatory liver function, including but not limited to total serum bilirubin (TBIL) above twice of the upper limit of normal (ULN), serum albumin (ALB) below 35 g/L or prothrombin activity (PTA) below 60% confirmed on repeated testing, previous or present history of ascites, upper gastrointestinal bleeding and/or hepatic encephalopathy, or with a liver function reserve of Child-Pugh class B or C.
* Primary liver cancer confirmed or evidenced by serum alfa-fetoprotein (AFP) above 100 ng/ml or liver imaging study showing suspected nodules.
* liver disease of a non-HCV etiology (e.g. alcoholic liver disease, nonalcoholic steatohepatitis, drug-induced hepatitis, autoimmune hepatitis, Wilson disease or hemochromatosis, etc.).
* Subjects has the following laboratory parameters at screening: ALT or AST>10×ULN, WBC < 3×109 /L, ANC< 1.5×109 /L（or < 1.25×109 /L for cirrhotics ), PLT< 50×109 /L, Hb < 100 g/L, INR > 1.5×ULN, CLcr < 50 mL/min（calculated by the Cockcroft-Gault equation ）.
* Uncontrolled diabetes mellitus (HbA1c > 8.0% at screening).
* Uncontrolled hyperthyroidism or diminished.
* Psychiatric or neurologic disorders, including previous or family history of psychiatric disorders (especially depression, depressive state, epilepsy or hysteria).
* Serious cardiovascular disorders, including uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥100 mmHg), heart insufficiency of New York Heart Association class III or above, history of myocardial infarction within 6 months before the screening, history of percutaneous transluminal coronary angioplasty within 6 months before the screening, unstable angina pectoris, or QTc interval (Fridericia correction formula QTc = QT×RR^-1/3) at or above 450 mse, second- or third-grade atrioventricular block or any other uncontrolled arrhythmias confirmed on repeated electrocardiography on screening.
* Serious hematologic disorders (e.g. anemia, hemophilia, etc.).
* Serious kidney diseases (e.g. chronic kidney disease, kidney insufficiency, etc.).
* Serious gastrointestinal disorders, (e.g. peptic ulcer, colitis, etc.) or post operative condition that could interfere with the absorption of the study drug.
* Serious respirator disorders, (e.g. active pulmonary tuberculosis, lung infection, chronic obstructive pulmonary disease, pulmonary interstitial disease, etc.).
* Malignancy within the 5 years prior to screening, with the exception of specific cancers that have been cured by surgical resection (basal cell skin cancer, etc).
* Solid organ transplantation.
* Hypersensitive predisposition or a known history of serious allergy, especially to the investigational products and substances.
* Positive urine drug screening at screening, or Clinically-relevant alcohol or drug abuse within 12 months of screening, and compliance and effectiveness evaluated by the investigator.
* Positive screening serum pregnancy test or baseline/day 1 serum or urine pregnancy test, and women are confirmed in pregnancy or lactation.
* Women of childbearing age (menopausal women aged ≤ 50 years old are also considered to have fertility), or partners who are women of childbearing age cannot comply with voluntary effective contraceptive measures during the 6 months from screening to the last dose of test drug.
* Use of any prohibited concomitant medications as described in protocol.
* Participated in clinical studies or previously participated within 3 months prior to baseline/Day 1.
* Conditions which investigator judges that it is not suitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2019-03-29 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Sustained virologic response at 12 weeks after end of treatment (SVR12) | 12 weeks after end of treatment
  Percentage of subjects with plasma HCV not detected or below the lower limit of quantitation (15 IU/mL)

SECONDARY OUTCOMES:
Rapid virologic response at 4 week after initiation of treatment (RVR4) | 4 week after initiation of treatment
  Percentage of subjects with plasma HCV not detected or below the lower limit of quantitation (15 IU/mL)
Rapid virologic response at 12 weeks after initiation of treatment (RVR12) | 12 weeks after initiation of treatment
  Percentage of subjects with plasma HCV not detected or below the lower limit of quantitation (15 IU/mL)
Sustained virologic response at 4 weeks after end of treatment (SVR4) | 4 weeks after end of treatment
  Percentage of subjects with plasma HCV not detected or below the lower limit of quantitation (15 IU/mL)
Sustained virologic response at 24 weeks after end of treatment (SVR24) | 24 weeks after end of treatment
  Percentage of subjects with plasma HCV not detected or below the lower limit of quantitation (15 IU/mL)
Virologic breakthrough | 2, 4, 8 and 12 weeks after initiation of treatment
  Percentage of subjects with on-treatment re-detected plasma HCV RNA after HCV RNA below the lower limit of quantitation
Virologic relapse | 4 and 12 weeks after end of treatment
  Percentage of subjects with off-treatment re-detected plasma HCV RNA after end-of-treatment HCV RNA below the lower limit of quantitation
Antiviral effects of SH229 tablets combined with Daclatasvi dihydrochloride (DCV) tablets , as measured by HCV RNA levels | Up to 36 weeks
  To evaluate the kinetics of circulating HCV RNA during treatment and after cessation of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Junqi Niu, Ph.D, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Jilin, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hua R, Kong F, Li G, Wen X, Zhang Y, Yang X, Meng C, Xie W, Jiang Y, Wang X, Han X, Huang Y, Mao Q, Wang J, Guan Y, Chen J, Ma Y, Xiong Q, Ma H, Yan X, Rao H, Zhao Y, Sun T, Zhu L, Mao X, Lian J, Deng G, Xin Y, Wang Y, Ye Y, Xu B, Gao H, Tan Y, Li D, Yang D, Su M, Zhang X, Min J, Shi X, Wei L, Niu J. Alfosbuvir plus Daclatasvir for Treatment of Chronic Hepatitis C Virus Infection in China. Infect Dis Ther. 2023 Nov;12(11):2595-2609. doi: 10.1007/s40121-023-00872-4. Epub 2023 Oct 19. PMID 37856013
- [Derived] Hua R, Kong F, Wen X, Xiong Q, Chen J, Meng C, Ma H, Tan Y, Huang Y, Jiang Y, Guan Y, Mao X, Wang J, Xin Y, Gao H, Xu B, Li C, Wu Q, Zhang X, Wang Z, Zhao L, Zhang Y, Li G, Niu J. Efficacy and safety of alfosbuvir plus daclatasvir in Chinese patients with hepatitis C virus genotypes 1, 2, 3, and 6 infection: An open-label, phase 2 study. J Viral Hepat. 2022 Jun;29(6):455-464. doi: 10.1111/jvh.13650. Epub 2022 Apr 8. PMID 35080256